CLINICAL TRIAL: NCT04588350
Title: Prospective, Multicenter, Single-arm Clinical Investigation Evaluating the Safety, Performance and Clinical Benefit of a New Autotransfusion Device in Cardiac Surgery
Brief Title: Clinical Investigation Evaluating a New Autotransfusion Device in Cardiac Surgery
Acronym: i-TRANSEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i-SEP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETC2017-002
Record Dates: First submitted 2020-09-28; First posted 2020-10-19 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Hemorrhage; Blood Loss; Surgical Blood Loss
Keywords: Autotransfusion; Cell salvage; Patient blood management
MeSH Terms: conditions — Hemorrhage; Blood Loss, Surgical

STUDY DESIGN:
Intervention Model Description: Single arm study in cardiac surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- i-SEP autotransfusion system (Experimental): Use of i-SEP autotransfusion system during the surgery
  Interventions: Device: i-SEP autotransfusion system

INTERVENTIONS:
Device: i-SEP autotransfusion system — Intraoperative recovery and washing of the processed blood by i-SEP autotransfusion system in surgeries where a bleeding is expected
  Other Names: same TM; MT0003; i-SEP ATS

SUMMARY:
Blood transfusion is at the heart of the therapeutic arsenal when there is a hemorrhage and/or blood loss during a surgery. There are two types of transfusion: the homologous one (blood from a compatible donor) and the autologous or autotransfusion method (which is done with the patient's own blood).

Although homologous transfusions can save lives, it can cause significant adverse events. Since then, multiple solutions have been developed to avoid exposing patients to these risks. It is in this context that was born the "Patient Blood Management" (PBM). Thus, the strategy in this PBM has been defined as "the appropriate use of blood and blood components, with the aim of minimizing the use of allogeneic transfusions".

In this context, particular interest has been given to autologous transfusion or autotransfusion or cell salvage, the general purpose is to reduce (or even stop) the use of allogeneic products and to reduce the risks associated with the ABO compatibility system, as well as all the adverse effects associated with allogeneic plasma and platelet transfusions.

Most autotransfusers available on the market operate by centrifugation. Autotransfusion is already a solution in Patient Blood Management and its efficiency and safety have already been optimized. However, there is still a need to improve the quality of the treated blood with an easier-to-use device that could improve the quality of the blood concentrate.

Indeed, with the current devices, it may happen that the use of allogeneic transfusions, plasma and platelets transfusions, is necessary in addition to autologous red blood cells thus reducing the interest of autotransfusion.

It is in this context that i-SEP has developed a new autotransfusion device based on a filtration method. Unlike competing devices, the i-SEP device allows the concentration of not only red blood cells (as competitive devices) but also platelets.

In this study, the i-SEP device is used in typical clinical applications of autotransfusion: cardiovascular and orthopedic surgeries, where there is a risk of hemorrhage and/or blood loss for example ≥ 500mL in cardiac surgery and ≥ 300mL in orthopedic surgery.

The study includes a screening phase (≤ 21Days), surgery phase when the i-SEP device is used (Day 0), a post-surgery phase (Day 1 - Day 6), a first follow-up visit (Day 7 ± 3) and a second follow-up visit (Day 30 ± 7).

DETAILED DESCRIPTION:
Blood transfusion is at the heart of the therapeutic arsenal when one wishes to preserve the hemodynamic balance of a patient. There are two types of transfusion: the homologous one (blood from a compatible donor) and the autologous or autotransfusion method (which is done with one's own blood / by the patient's own blood).

Although homologous transfusions can save lives, it may lead to non-negligible adverse events. Among these events, immunological consequences such as allo-immunization against red blood cells' antigens from the donor blood can be cited. Some infections have also been reported following allogenic transfusions.

Since then, multiple solutions have been developed to avoid exposing patients to these risks. It is in this context that was born the "Patient Blood Management" (PBM). Thus, the strategy in this PBM has been defined as "the appropriate use of blood and blood components, with the aim of minimizing the use of allogeneic transfusions". In this context, particular interest has been given to autologous transfusion or autotransfusion or cell salvage.

The principle of Intra-Operative Cell Salvaged (IOCS) allows intravenous administration of the patient's own blood collected at the surgical site or postoperative wound during hemorrhagic surgery. It is used mainly in cardiac, vascular, transplant and elective orthopedic surgeries and tends to spread to other surgeries such as neurosurgery, obstetrics and urology.The IOCS has multiple benefits, primarily autologous (the patient gets his own blood), immediate availability in the operating room, reduced costs of patient care, and the recycling of otherwise lost blood products. It is part of blood saving techniques that avoid the use of homologous blood. Indeed, the general purpose of IOCS is to reduce (or even stop) the use of allogeneic products and to reduce the risks associated with the ABO compatibility system, as well as all the adverse effects associated with allogeneic plasma and platelet transfusions

Most autotransfusers available on the market operate by centrifugation. Autotransfusion is already a solution in Patient Blood Management and its efficiency and safety have already been optimized. However, there is still a need to improve the quality of the treated blood with an easier-to-use device that could improve the quality of the blood concentrate.

Indeed, with the current devices, it may happen that the use of allogeneic transfusions, plasma and platelets transfusions, is necessary in addition to autologous red blood cells thus reducing the interest of autotransfusion.

It is in this context that i-SEP has developed a new autotransfusion device based on a filtration method. Unlike competing devices, the i-SEP device allows the concentration of not only red blood cells (as competitive devices) but also platelets.

In this study, the i-SEP device is used in typical clinical applications of autotransfusion: cardiovascular and orthopedic surgeries, where there is a risk of hemorrhage and/or blood loss for example ≥ 500mL in cardiac surgery and ≥ 300mL in orthopedic surgery.

The study includes a screening phase (≤ 21Days), surgery phase when the i-SEP device is used (Day 0), a post-surgery phase (Day 1 - Day 6), a first follow-up visit (Day 7 ± 3) and a second follow-up visit (Day 30 ± 7).

ELIGIBILITY:
Inclusion Criteria:

Preoperative Inclusion Criteria:

* Is the patient able and willing to give informed consent before participating in the study?
* Is the patient aged ≥ 18 years?
* Does the patient have a social protection system?
* Does the patient weigh ≥ 59kg (for the sole purpose of blood assessment related to the clinical study)?
* Is the patient indicated for a cardiac surgery with the implementation of a Cardio Pulmonary Bypass (CPB)?
* Does the patient have a preoperative hemoglobin ≥ 13g / L for a man and ≥ 12g / L for a woman?
* Does the patient have a preoperative platelets count ≥ 150000 / μL?

Intraoperative Inclusion Criteria:

- Does the patient have anticoagulated blood losses ≥ 500mL (without considering priming volume in the first cycle)?

Exclusion Criteria:

Preoperative Exclusion Criteria:

* Is the patient indicated for a surgery because of a suspected or confirmed cancer?
* Does the patient have any systemic or local infection in the area of intervention, suspected or proven?
* Does the patient have any pathology of hemostasis (Hemophilia, ...) or bleeding disorder confirmed, or strongly suspected on the examination of the patient in consultation (high score on the formalized questionnaire: HEMSTOP)?
* Is the patient's life expectancy of less than 2 months?
* Does the patient have any psychiatric condition that could, in the opinion of the investigator, prevent him / her from participating in this study?
* Does the patient have any objections to transfusion (homologous)?
* Is the patient participating in or has participated in another clinical study in the last 30 days at the day of screening and has received (or is receiving) treatments that could have an impact on the effectiveness of the autotransfusion?
* Does the investigator consider that the patient (or the surgical conditions) is not appropriate to be included in this clinical study?
* Does the patient have a TIH - Heparin-Induced Thrombocytopenia - suspected or confirmed and therefore cannot receive heparin?
* Is the patient pregnant or a lactating woman?
* Is the patient a woman of childbearing age who is not on effective contraceptive treatment?
* Is the patient due to have combined surgeries?
* Has the patient been admitted for an emergency surgery?
* Does the patient have an endocarditis?
* Has the patient been admitted for a redux surgery?
* Has the patient been admitted for a heart transplantation or a mechanical circulatory support surgery?
* Has the patient been admitted for congenital heart surgery?
* Has the patient taken

  * any anti-platelet aggregation drugs (except acid acetylsalicylic - aspirin) including Ticagrelor, Clopidogrel and Prasugrel or,
  * any anticoagulant drugs (intake of vitamin K antagonists or DOAC = direct oral anti-coagulant including rivaroxaban, Edoxaban, Apixaban and Dabigatran), outside the recommendations from EACTS / EACTA and GHIP?

Intraoperative Exclusion Criteria:

- Is the "emergency" mode available on the i-Sep machine used during surgery?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Safety of the device in terms of elimination of contaminants such as heparin and hemolysis markers (free hemoglobin) | Day 0
  Proportion of patients with heparin washout ≥ 90% and with free hemoglobin washout ≥ 75% on the concentrated blood from the i-SEP device
Performance of the device in terms of exceeding red blood cell recovery and hematocrit / hemoglobin thresholds | Day 0
  Proportion of patients with mean Red Blood Cells (RBCs) recovery ≥ 80% and with mean output Hematocrit ≥ 40% or hemoglobin concentration ≥ 13.3g/dL. Mean recovery is calculated with quantification in the pre-treatment blood (after pre-filtration through the blood collection reservoir) and quantification in the concentrated blood, mean output is calculated on the concentrated blood.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 1 month follow-up
  Proportion of patients with adverse events (especially Serious Adverse Events, Serious Adverse Device Effects)
Incidence of homologous transfusion | Up to 1 month follow-up
  Proportion of patients with homologous transfusion (number of units and type of blood product infused) during operative and post-operative period
Incidence of re-intervention for bleeding | Up to 1 month follow-up
  Proportion of patients with re-intervention for bleeding during post-operative period
Contaminants concentration such as heparin and hemolysis markers (free hemoglobin) in the concentrated blood | Day 0
  Concentration of heparin and free hemoglobin in the treated (concentrated) blood from the i-SEP device
Evolution of the patient's complete blood count | Up to Day 2
  Evolution of the patient complete blood count after surgery as compared to before surgery
Blood loss in drainage after surgery | Up to Day 2 and/or to drainage removal
  Quantity and evolution of the patient blood loss in drainage after surgery
White Blood Cells yield | Day 0
  Quantification of White Blood Cells in the pre-treatment blood (after pre-filtration through the blood collection reservoir) and in the concentrated blood from the i-SEP device
Hematocrit yield | Day 0
  Quantification of hematocrit in the pre-treatment blood (after pre-filtration through the blood collection reservoir) and in the concentrated blood from the i-SEP device
Hemoglobin yield | Day 0
  Quantification of hemoglobin in the pre-treatment blood (after pre-filtration through the blood collection reservoir) and in the concentrated blood from the i-SEP device
Total protein yield | Day 0
  Quantification of total protein in the pre-treatment blood (after pre-filtration through the blood collection reservoir) and in the concentrated blood from the i-SEP device
Albumin yield | Day 0
  Quantification of albumin in the pre-treatment blood (after pre-filtration through the blood collection reservoir) and in the concentrated blood from the i-SEP device
Potassium yield | Day 0
  Quantification of potassium in the pre-treatment blood (after pre-filtration through the blood collection reservoir) and in the concentrated blood from the i-SEP device
Fat yield through triglyceride assay | Day 0
  Quantification of fat through triglyceride measurements in the pre-treatment blood (after pre-filtration through the blood collection reservoir) and in the concentrated blood from the i-SEP device
Performance of the device in terms of platelets recovery | Day 0
  Platelet yield and their functionality through platelet activation and degranulation measured in the pre-treatment blood (after pre-filtration through the blood collection reservoir) and in the concentrated blood from the i-SEP device
High levels of red blood cell recovery and hematocrit / hemoglobin thresholds | Day 0
  Proportion of patients with mean output Hematocrit ≥ 45% or hemoglobin concentration ≥ 15.5g/dL in the concentrated blood from the i-SEP device

OTHER OUTCOMES:
User satisfaction questionnaire | Through study completion, an average of 1 year
  Each user fills in a questionnaire to give its feeling about the ergonomics and intuitivity of the i-Sep device

CONTACTS AND LOCATIONS:
Overall Officials: Francis Gadrat, MD, Study Chair — i-SEP; Nicolas Nesseler, MD, Principal Investigator — CHU de Rennes, Rennes, France
Locations (5):
- France (5):
  - CHU de Bordeaux - GH Pellegrin, Bordeaux
  - CHU de Nantes, Nantes
  - Ap-Hp - Hegp, Paris
  - CHU de Bordeaux - GH Sud, Pessac
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mansour A, Beurton A, Godier A, Rozec B, Zlotnik D, Nedelec F, Gaussem P, Fiore M, Boissier E, Nesseler N, Ouattara A. Combined Platelet and Red Blood Cell Recovery during On-pump Cardiac Surgery Using same by i-SEP Autotransfusion Device: A First-in-human Noncomparative Study (i-TRANSEP Study). Anesthesiology. 2023 Sep 1;139(3):287-297. doi: 10.1097/ALN.0000000000004642. PMID 37294939